CLINICAL TRIAL: NCT05616286
Title: Mindfulness-SOS for Refugees: Randomized Controlled Trial
Brief Title: Mindfulness-SOS for Refugees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Mindfulness-SOS RCT
Record Dates: First submitted 2022-11-06; First posted 2022-11-15 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-09

CONDITIONS: Stress Disorders, Post-Traumatic; Stress Related Disorder
Keywords: Forcibly Displaced Persons; Post-Migration Stress; Trauma; Depression; Anxiety; Stress; Online Mental Health Intervention Program; Mindfulness; Compassion; Treatment Adherence
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries; Depression; Anxiety Disorders; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-SOS (Experimental): Mindfulness-SOS for Refugees is a brief internet-based mobile-supported intervention program which is a mobile health adaptation of MBTR-R, mindfulness- and compassion-based, trauma-sensitive, and socio-culturally adapted group intervention program designed for FDPs. Mindfulness-SOS for Refugees entails 8 brief sessions and 9 mindfulness meditation practice exercises - delivered via audio recordings using participants' smartphones. Mid-intervention, 3-weeks following randomization, all participants will be re-assessed. Participants initially randomized to MG-Mindfulness-SOS will be identified as either responders or non-responders. Responders will be assigned to continue MG-Mindfulness-SOS. Non-responders will be re-randomized to either Intensified-Guidance Mindfulness-SOS (IG-Mindfulness-SOS), an adaptive intervention sequence condition, or to continue with the MG-Mindfulness-SOS, a non-adaptive intervention sequence condition.
  Interventions: Behavioral: Mindfulness-SOS for Refugees
- Waitlist-Control (No Intervention): Following the 7-week waitlist period and another assessment, participants randomized to waitlist-control will be assigned to Minimally-Guided Mindfulness-SOS (MG-Mindfulness-SOS) and then re-assessed following 3-weeks and, as described above, assigned to either continue in the MG-Mindfulness-SOS group or to move to the Intensified-Guidance Mindfulness-SOS (IG-Mindfulness-SOS).

INTERVENTIONS:
Behavioral: Mindfulness-SOS for Refugees — Mindfulness-SOS for Refugees is a brief internet-based mobile-supported intervention program which is a mobile health adaptation of MBTR-R, mindfulness- and compassion-based, trauma-sensitive, and socio-culturally adapted group intervention program designed for FDPs. Mindfulness-SOS for Refugees entails 8 brief sessions and 9 mindfulness meditation practice exercises - delivered via audio recordings using participants' smartphones. The Mindfulness-SOS for Refugees intervention program is specifically designed to mitigate acute stress and related mental health symptoms among FDPs.
  Arms: Mindfulness-SOS

SUMMARY:
Worldwide, refugees and asylum seekers suffer at high rates from trauma and stress-related mental health problems. The research group therefore developed, and initially piloted in a single-site open trial, a novel mindfulness- and compassion-based digital intervention program - Mindfulness-SOS for refugees (Mindfulness-SOS). The pilot study had promising preliminary findings of utilization, feasibility and related dose-response effects of intervention program engagement with mental health outcomes. The digital intervention program was developed based on randomized control trial data of a group-based mindfulness- and compassion-based program for forcibly displaced people.

To address common limitations of mobile health interventions such as attrition, engagement and adherence, the investigators will implement a personalized stepped-care adaptation and augmentation of Mindfulness-SOS, that entails providing intensified (remote) guidance for FDPs that do not respond to the intervention, to optimize capacity to therapeutically benefit from Mindfulness-SOS. To do so, the investigators propose to carry out a randomized controlled Sequential Multiple Assignment Randomized Trial (SMART) study to test and optimize the therapeutic outcomes of Mindfulness-SOS, using an adaptive intervention sequence of guidance format intensities among N ≅ 170 (50% female) adult trauma-affected Eritrean asylum-seekers residing in Israel.

DETAILED DESCRIPTION:
Over 100 million Forcibly Displaced Persons (FDPs), including refugees and asylum-seekers, are forcibly displaced due to conflict, persecution, and natural disaster. Forced displacement is often associated with severe and chronic forms of trauma- and stress-related mental health difficulties, with destructive generational and inter-generational consequences for forcibly displaced families including spouses or partners, children, as well as communities.

To address this fast-growing crisis and the public health challenge, field-wide efforts have emerged to develop and test interventions tailored to the complex needs and post-displacement settings of FDPs. Among such efforts, the research group developed Mindfulness-Based Trauma Recovery for Refugees (MBTR-R) - a Mindfulness-Based Intervention (MBI) that is group-based, trauma-sensitive and socio-culturally adapted for diverse populations of FDPs. MBTR-R demonstrated waitlist-controlled evidence of efficacy and safety to improve stress- and trauma-related mental health outcomes among African asylum-seekers in Israel.

Yet, the potential reach, access, scalability, and therefore impact of such interventions is systematically limited by their relatively rigid, group-based in-person delivery format. Behavioral Intervention Technologies (BITs), notably via mobile health interventions (mHealth), may be one promising implementation approach to help facilitate the dissemination and scalability of MBTR-R among FDPs. The research group therefore developed, and initially piloted a novel mHealth adaptation of MBTR-R - Mindfulness-SOS for refugees (Mindfulness-SOS) with promising preliminary findings of utilization, related feasibility and effects of engagement with the program on several individual mental health outcomes (i.e., modest protective dose-response effects).

Yet, to improve their impact and efficacy, the development and delivery of BIT adaptations of MBIs broadly, and among FDPs specifically, must address well-documented limitations of BITs, most notably, high attrition, low engagement and adherence. One way to do so is through personalized stepped-care adaptation and augmentation of Mindfulness-SOS, that entails providing intensified (remote) guidance for FDPs that do not respond to the intervention, as a means of reducing attrition, increasing engagement and adherence, and optimizing capacity to therapeutically benefit from Mindfulness-SOS. The research group argues that a Sequential Multiple Assignment Randomized Trial (SMART), a multistage randomized trials design, is particularly well-suited to experimentally deliver, test, and optimize such a personalized adaptive stepped-care approach to Mindfulness-SOS for FDPs.

The research group therefore propose to carry out a SMART study to test and optimize the therapeutic outcomes of Mindfulness-SOS, using an adaptive intervention sequence of guidance format intensities among N ≅ 170 (50% female) adult Eritrean asylum-seekers residing in Israel. Following baseline assessment (pre-intervention), participants will be randomly assigned to Minimally-Guided Mindfulness-SOS (MG-Mindfulness-SOS) or to Wait-List Control. Mid-intervention, 3-weeks following randomization, all participants will be re-assessed. Participants initially randomized to MG-Mindfulness-SOS will be identified as either responders or non-responders. Responders will be assigned to continue MG-Mindfulness-SOS. Non-responders will be re-randomized to either Intensified-Guidance Mindfulness-SOS (IG-Mindfulness-SOS), an adaptive intervention sequence condition, or to continue with the MG-Mindfulness-SOS, a non-adaptive intervention sequence condition. Following the 7-week wait-list period and after re-assessment, Wait-List Control participants will initiate MG-Mindfulness-SOS intervention, receive MG-Mindfulness-SOS. Then, like participants initially randomized to MG-Mindfulness-SOS, 3-weeks following the wait-list period, participants will be re-randomized to either Intensified-Guidance Mindfulness-SOS (IG-Mindfulness-SOS), the adaptive intervention sequence condition, or to continue with the MG-Mindfulness-SOS, the non-adaptive intervention sequence condition. All participants will be re-assessed at post-intervention, and then at 8-week follow-up assessment. Primary outcomes will include subjective self-report measures of individual mental health outcomes. Secondary outcomes will include subjective self-report and/or parental report measures of pro-social family outcomes, child outcomes, inter-personal and community outcomes.

ELIGIBILITY:
Inclusion Criteria:

* East African refugee or asylum seeker living in Israel
* Tigrinya fluency and literacy
* Owns a personal smartphone

Exclusion Criteria:

* Active suicidal ideation or/and past suicide attempt in the last year or/and passive suicidal ideation with clinical indicators of imminent suicide risk (e.g. severe paranoia)
* Current mental health treatment (i.e. psychotherapy or/and group therapy at least twice a month)
* Participation in the MBTR-R group in a previous study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Harvard Trauma Questionnaire | Change from immediately pre-intervention to 1-week post-intervention
  The Harvard Trauma Questionnaire (HTQ) is a 16-item self-report questionnaire to assess post-traumatic stress symptom severity (5-point Likert scale) with higher scores indicating greater post-traumatic stress severity (minimum scale score 1 and maximum scale score 5), HTQ mean cut-off score ≥ 2 is commonly used to identify categorical (diagnostic) symptom status of post-traumatic stress disorder
Brief Patient Health Questionnaire (PHQ-9) | Change from immediately pre-intervention to 1-week post-intervention
  A 9-item self-report questionnaire to assess depression symptom severity (5-point Likert scale) with higher scores indicating greater depression symptom severity (minimum scale score 0 and maximum scale score 36), PHQ-9 mean cut-off score ≥10 is commonly used to identify categorical (diagnostic) symptom status of depression.
Beck's Anxiety Inventory (BAI) | Change from immediately pre-intervention to 1-week post-intervention
  The Beck's Anxiety Inventory (BAI) is a 21-item self-report questionnaire to assess anxiety symptom severity (4-point Likert scale) with higher scores indicating greater anxiety symptom severity (minimum scale score 0 and maximum scale score 63), BAI total cut-off score ≥ 16 is commonly used to identify categorical (diagnostic) symptom status of anxiety disorder.
Positive and Negative Affect Schedule (PANAS) | Change from immediately pre-intervention to mid-assessment (3 weeks in) to 1-week post-intervention
  PANAS-SF is a 10-item self-report questionnaire measuring state positive and negative affect (5-point Likert scale ranging from 1 to 5) with higher scores indicating greater state positive and negative affect. The PANAS-SF includes 2 subscales, one measuring positive affect and the other measuring negative affect. Each subscale score is the sum of its items.

SECONDARY OUTCOMES:
Post-Migration Living Difficulties (PMLD) scale | Change from immediately pre-intervention to 1-week post-intervention
  The Post-Migration-Living-Difficulties Checklist (PMLD) is a 9-item self-report questionnaire to assess post-migration stress (5-point Likert scale) with higher scores indicating greater post-migration stress (minimum scale score 1 and maximum scale score 5).
Brief Inventory of Thriving (BIT) | Change from immediately pre-intervention to 1-week post-intervention
  One item of the 9-item self-report questionnaire Brief Inventory of Thriving (BIT) was used to assess subjective wellbeing (5-point Likert scale) with higher scores indicating greater subjective well-being (minimum score 1 and maximum score 5).
The State Shame and Guilt Scale | Change from immediately pre-intervention to 1-week post-intervention
  The State Shame and Guilt Scale (SSGS) is a 15-item self-report questionnaire to assess state shame and guilt (5- point Likert scale) with higher scores indicating greater levels of state shame, guilt and pride (minimum scale score 15 and maximum scale score 75).
Brief Five-Facet-Mindfulness Scale | Change from immediately pre-intervention to 1-week post-intervention
  The Five Facets of Mindfulness Questionnaire (FFMQ) is a self-report questionnaire to assess different facets of trait mindfulness (5-point Likert scale) with higher scores indicating greater levels of trait mindfulness (minimum scale score 1 and maximum scale score 5).
Short Form of the Conflict Tactic Scale | Change from immediately pre-intervention to 1-week post-intervention
  The Conflict Tactics Scales (CTS2) is the most widely used instrument for measuring intimate partner violence. The scale presents various cases of intimate partner violence and measures the frequency of these instances. The scale consists of 16 items measured on a 5-point scale ranging from (1)This has never happened to (5) 3-5 times in the last week.
Revised Social Capital Scale | Change from immediately pre-intervention to 1-week post-intervention
  The social capital scale is used to measure the resources available to an individual through relational networks. The scale consists of 11 items on a 5-point Likert scale ( 1- Not at all - 5-Very often).
Sussex-Oxford Compassion for Self Scale | Change from immediately pre-intervention to 1-week post-intervention
  The Self-Compassion Scale SOCS is a 20-item self-report questionnaire to assess different facets of compassion for others (5-point Likert scale) with higher scores indicating greater levels of compassion for others (minimum scale score 1 and maximum scale score 5).
Challenged Sense of Belonging Scale (CSBS) | Change from immediately pre-intervention to 1-week post-intervention
  The CSBS assess a challenged or eroded sense of belonging that provides insight into how individuals relate to their environment and how socially connected they feel. The scale consists of four key elements connection, participation, identification, and congruence. The CSBS is a 4-item scale measured in a 5-point Likert scale ranging from 1(Strongly agree)-5(Strongly disagree).
Metacognitive Processes of Decentering Scale-Trait (MPoD-T) | Change from immediately pre-intervention to 1-week post-intervention
  MPod-s is a 3-item self-report questionnaire measuring state levels of the 3 metacognitive processes of decentering (11-point Likert scale ranging from 0 to 10) with higher scores indicating greater levels of decentering (minimum scale score 0 and maximum scale score 10). Each of the 3 MPoD-s items measures a metacognitive process of decentering: meta-awareness, disidentification from internal experience, and non-reactivity to internal experience. MPod-s will be used to measure change, from pre-to post-intervention, instate decentering during the MAT mindfulness meditation.
Alliance with an Unguided Smartphone App | Change from immediately pre-intervention to 1-week post-intervention
  The measure consists of 6 items on a 5-point Likert scale 1(strongly agree)-5(strongly disagree). The measure aims to determine the quality of the alliance between the app-user and the smartphone app.
Child Behavior Checklist (CBCL) | Change from immediately pre-intervention to 1-week post-intervention
  The CBCL includes 21 items measured on a 3-point Likert scale (0-Never true - 2-Often true). The measure is used to detect behavioral and emotional problems in children and adolescents.
Hostile/Warm Parenting styles | Change from immediately pre-intervention to 1-week post-intervention
  This measure consists of items that measure parental warmth and parental hostility. The measure consists of 11 items on a 5-point Likert scale 1(never)-5(always).
Brief Problem monitoring (BPM) | Change from immediately pre-intervention to 1-week post-intervention
  The BPM provides a uniformed problem scale to assess attentional, behavioral, and internalizing problems in children and adolescents aged from 6-18 years old. The BPM includes 19 items measured on a 3-point Likert scale (0-Not true - 2-Very true).

CONTACTS AND LOCATIONS:
Locations (1):
- Central Bus Station, Tel Aviv, Israel